CLINICAL TRIAL: NCT05138185
Title: Evaluation of the Effects of the Unilateral Assistance Provided by a Robotic Knee Exoskeleton in the Gait Symmetry of Healthy Subjects and Hemiparetic Patients.
Brief Title: Proof-of-concept of a Robotic Knee Exoskeleton in Healthy Subjects and Hemiparetic Patients During Gait.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish National Research Council (Other Government)
Collaborators: Hospital Beata María Ana (Other)
Responsible Party: Principal Investigator, Julio S. Lora Millan, Responsible Engineer, Spanish National Research Council
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: REFLEX_TechValidation
Record Dates: First submitted 2021-10-23; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Hemiparesis/Hemiplegia (One Sided Weakness/Paralysis)
Keywords: Hemiparetic Gait; Robotic Knee Exoskeleton
MeSH Terms: conditions — Paresis; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Exoskeleton assisted gait on a treadmill — Subjects were instructed to walk on a treadmill at a constant speed during trials of 5 minutes. All subjects carried out four trials: (1) NoExo: subjects only wore the sensors to acquire their basal motion; (2) Free: subjects wore the exoskeleton although the actuator was mechanically decoupled, so it enabled the free movement of the knee; (3) Echo: the device provided gait assistance following the Echo-control strategy; and (4) Pattern: the device provided gait assistance following the Pattern strategy. During trials, patients wore a safety harness that did not support any weight. Previously to the execution of the trials, the gait velocity was self-selected by the subjects to a comfortable level. Subjects rested between trials for five minutes. Healthy subjects also performed a previous trial under variable gait speed. They walked over the treadmill as in the NoExo condition, although the gait speed randomly varies from 1km/h to 3km/h in 0.2km/h steps for 15 seconds at least.

SUMMARY:
Hemiparetic gait is characterized by strong asymmetries that could severely affect the quality of life of stroke survivors. This asymmetry is due to motor deficits in the paretic leg and the resulting compensations in the non-paretic limb.

In this study, the investigators aim to evaluate the effect of actively promoting gait symmetry in hemiparetic patients by assessing the behavior of both paretic and non-paretic lower limbs. To this end, the investigators use a unilateral active Knee-Ankle-Foot Orthosis able to assist the paretic limb of hemiparetic patients during gait.

The system is able to synchronize its action with the movement of the unassisted joints, promoting a natural and intuitive interaction. The device generate the assistance according to two differents strategies: (1) Replicating the movement of the helathy leg or (2) Inducing a healthy gait pattern on the paretic leg.

The hypothesis is that a proper and natural interaction between the user and the exoskeleton would enable the patients to consider the robot action as a part of their own gait capability, improving their gait quality as consequence. Hemiparetic asymmetry is not only due to impairments in the affected limb, but also it is the consequence of biomechanical compensatory mechanisms that might arose in the non-paretic leg. We aim to assess the adaptation process of the subject to the exoskeleton assistance, and to evaluate the effects of such human-robot interaction in both paretic and non-paretic legs.

DETAILED DESCRIPTION:
- Brief name: Proof-of-concept of a unilateral robotic knee exoskeleton and evaluation of its effects over gait symmetry.

- Materials: The investigators have developed a Knee-Ankle-Foot orthosis (KAFO) composed of two joints aligned to the knee and ankle of the user. The length of its bars and the positions of its braces can be tailored to the anthropometry of different users. The knee joint is actuated by a DC brushless motor EC-60 flat 408057 (Maxon ag, Switzerland) coupled with a harmonic drive CSD-20-160-2AGR (Harmonic Drive LLC, EE.UU.). The transmission ratio of 1:60 of this system enables the application of a mean torque of 35Nm. The ankle joint of the prototype remains non-actuated and unlimited, enabling its free movement in the sagittal plane. The total weight of the KAFO is about 4kg.

The prototype is equipped with sensors that provide information on system variables that are used for its control in real-time, such as the flexion angle of the robot joint or the interaction torque between user and robot. In addition, the gait kinematic of the user is measured by Inertial Measurement Units (IMUs) and the contact of both feet with the floor by Force Sensing Resistors (FSRs).

The system uses an Adaptive Frequency Oscillator to estimate the continuous gait phase of the contralateral limb and synchronically assists the paretic leg following two different control strategies: (1) Replicating the movement of the sound leg (Echo Strategy) or (2) Inducing a healthy gait pattern on the paretic leg (Pattern strategy). The action of the robot depends on the gait phase of the assisted leg: during stance the robot reinforces the limb so the system composed of the leg and the exoskeleton can load the user's weight and not collapse, while during the swing phase the robot guides the limb's movement according to the Assisted-As-Needed (AAN) paradigm creating a force tunnel around the prescribed trajectory.

- Procedures: Subjects were instructed to walk on a treadmill at a constant speed during trials of 5 minutes. All subjects carried out four different kinds of trials: (1) NoExo: subjects only wore the inertial sensors and the insole pressure sensors to acquire their basal motion; (2) Free: subjects wore the exoskeleton although the actuator was mechanically decoupled, so it enabled the free movement of the knee; (3) Echo: the device provided gait assistance following the Echo-control strategy; and (4) Pattern: the device provided gait assistance following the Pattern strategy. During trials, patients wore a safety harness, although it did not support any weight. Previously to the execution of the trials, the gait velocity was self-selected by the subjects to a comfortable level. Subjects rested between trials for five minutes at least, in order to avoid adaptation and learning effects from trial to trial.

Healthy subjects also performed a previous trial under variable gait speed (VariableSpeed). They walked over the treadmill as in the NoExo condition, although the gait speed randomly varies from 1km/h to 3km/h in 0.2km/h steps for 15 seconds at least.

- Intervention providers A physiotherapist and an engineer are present during the trials. The first is responsible of assessing the basal gait of the subjects and evaluating his/her state while the assistance is provided. The engineer is responsible of managing the device and recording the data.

Both researchers monitor fidelity to the intervention by direct supervision.

* Modes of delivery The protocol is provided to one participant at a time. Each patient completes the protocol once.
* Location Hospital Beata María Ana (Madrid, Spain)
* Tailoring and modifications The protocol remains unaltered across applications. The only adaptation to patients is the choice of the comfortable gait speed for the trials.

ELIGIBILITY:
Inclusion Criteria: Ischemic or hemorragic stroke that lead to hemiplegic gait or healthy subjects without gait impairements. Same number os subjects is recruited

Exclusion Criteria:

1. Acute musculoskeletal diseases
2. Peripheral vascular diseases
3. Acute cardiopulmonary diseases
4. Acute neurological diseases
5. Excessive spasticity in any joint of the lower limb (Ashworth scale> 2)
6. Joint mobility restriction of lower limb joints due to any cause
7. Pain due to impaired mobility of the lower limb
8. Inability to use robotic exoskeleton prototypes due to his/her health condition.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of the prototype device | During the last two minutes of the intervention
  The joints motion is measured by Inertial Sensors

SECONDARY OUTCOMES:
Symmetry of step length from thigh and shank kinematics | During the last two minutes of the intervention
  The joint motion is measured by Inertial Sensors
Symmetry of step time | During the last two minutes of the intervention
  Data is collected from floor contact events detected by FSRs

CONTACTS AND LOCATIONS:
Overall Officials: Julio S. Lora-Millan, Principal Investigator — Spanish National Research Council
Locations (1):
- Hospital Beata María Ana, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: Immediately following publication, no end date
Access Criteria: Access will be subject to methodologically sound proposals and it will be approval by scientific investigator (julio.lora@csic.es)